CLINICAL TRIAL: NCT05979155
Title: A Multicenter, Non-randomized, Open-label, Multiple-Dose Phase I Study of NWY001, in Subjects With Advanced Solid Tumors
Brief Title: A Study of NWY001 in Subjects With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NWY001-101
Record Dates: First submitted 2023-07-20; First posted 2023-08-07 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study arm (multiple doses of NWY001) (Experimental): Part 1: dose-escalation of monotherapy NWY001
  Interventions: Biological: NWY001
- Study arm (RP2D of NWY001) (Experimental): Part 2: dose-expansion of monotherapy NWY001
  Interventions: Biological: NWY001

INTERVENTIONS:
Biological: NWY001 — Part 1: Participants will be given a single-dose of NWY001 intravenously once every 3 weeks until a discontinuation criteria was met during treatment period.
  Arms: Study arm (multiple doses of NWY001)
Biological: NWY001 — Part 2: Participants will be given RP2D of NWY001 intravenously once every 3 weeks until a discontinuation criteria was met during treatment period.
  Arms: Study arm (RP2D of NWY001)

SUMMARY:
This is a Phase 1, single-arm, open-label, dose-escalation study in patients with advanced solid tumors including 2 parts:

Part 1: Dose-Escalation Part Part 2: Dose-Expansion Part

DETAILED DESCRIPTION:
Part 1: Patients with advanced solid tumors that has relapsed from or is refractory to standard therapy or for which no standard therapy exists will be enrolled in different cohorts.

Part 2: Recommended Phase 2 dose (RP2D) of NWY001 will be given to all patients enrolled in this part.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to sign a written informed consent document
2. Participant with advanced solid malignant tumor that has relapsed from or is refractory to standard therapy or for which no standard therapy exists
3. 18~75 years of age at the time of screening
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
5. Life expectancy ≥3 months
6. Laboratory tests meet the following criteria (no corrective treatment, such as G-CSF, erythropoietin, and blood transfusion, within 14 days before first dose):

1) absolute neutrophil count (ANC) ≥1.5×109/L 2) platelet ≥100×109/L 3) hemoglobin ≥90 g/L 4) creatinine clearance >50 mL/min (according to Cockcroft-Gault equation) 5) both alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤1.5×upper limit of normal (ULN) (≤5×ULN for patients with hepatic metastasis) 6) total bilirubin ≤1.5×ULN (≤3×ULN for patients with gilbert syndrome) 7) international normalized ratio (INR) <2.0, activated partial thromboplastin time (aPTT) ≤1.5×ULN

7. Prior anti-cancer therapy meets the following criteria:

1. major surgery ≥4 weeks
2. radiotherapy ≥4 weeks
3. endocrine therapy ≥2 weeks
4. chemotherapy (including antibody) ≥3 weeks
5. immunotherapy ≥4 weeks

8. At least one measurable target lesion as defined by RECIST1.1

9. For part 2a: Participant has a diagnosis of histologically confirmed advanced (unresectable) or metastatic gastric or gastroesophageal junction adenocarcinoma

1. participant with HER2 overexpression (IHC 3+ or IHC 2+/ISH+) is refractory or intolerant to standard therapy or for which no standard therapy exists. Prior treatment with trastuzumab or HER2-targeted drugs
2. participant with no HER2 expression is refractory or intolerant to standard therapy or for which no standard therapy exists

10. For part 2b: Participant has a diagnosis of histologically confirmed advanced esophageal squamous carcinoma

11. For part 2c: Participant has a diagnosis of histologically confirmed advanced pancreatic ductal adenocarcinoma

12. For part 2d: Participant has a diagnosis of histologically confirmed advanced hepatocellular carcinoma

13. For part 2e: Participant has a diagnosis of histologically confirmed advanced intrahepatic cholangiocarcinoma

14. For part 2f: Participant has a diagnosis of histologically confirmed advanced MSI-H/dMMR colorectal cancer

Exclusion Criteria:

1. Current or previous history of other active aggressive malignancies in the last 5 years, except :

1. previous history of non-aggressive malignancies, such as cervical carcinoma in situ, melanoma in situ, or ductal carcinoma in situ of the breast that remains in complete remission for years after curative treatment
2. malignancies with negligible risk of metastasis or death (such as adequately treated basal or squamous cell skin cancer and focal prostate cancer)

2. Current or previous history of hematological malignancies

3. Primary central nervous system (CNS) malignancies or CNS metastases

4. History of allergy or hypersensitivity to monoclonal antibodies or excipients, or a known history of allergy to antibodies produced by Chinese hamster ovary cell

5. Uncontrolled infection that requires intravenous antibiotics, antivirals, or antifungal medications

6. History of clinically significant lung diseases (such as interstitial pneumonia, pneumonia, pulmonary fibrosis, and severe radiation pneumonia), or patients suspected of having these diseases on radiographic examination during the screening period

7. Uncontrolled complications, including, but not limited to, persistent active infections, active coagulopathy, uncontrolled cardiovascular disease, uncontrolled immune disease, uncontrolled diabetes, uncontrolled chest and abdominal fluid accumulation, psychiatric disorders that do not meet study requirements, and other serious conditions requiring systemic treatment

8. Known history of HIV, active infections of hepatitis B or hepatitis C

9. Active pulmonary tuberculosis. Participants vaccinated with BCG vaccine may be false positive for PPD, and they could be enrolled if negative for IGRA

10. Women who are pregnant or breastfeeding or intended to become pregnant during the study period

11. Participants of childbearing potential who refuse to take highly effective contraceptive measures during the entire study treatment period and for 120 days after the last dose of study drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Up to 21 days
  Number of patients experienced any dose limited toxicity
Incidence of adverse events (AEs) | Until 30 days after the last dose of the study drug
  Number of patients experienced AEs

SECONDARY OUTCOMES:
Objective response rate (ORR) | Until 30 days after the last dose of the study drug
  The proportion of patients who have a complete response (CR) or partial response (PR), as determined by the Investigator at local site per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1
Disease control rate (DCR) | Until 30 days after the last dose of the study drug
  The proportion of patients who have a CR or PR or stable disease (SD), as determined by the Investigator at local site per RECIST 1.1
Progression free survival (PFS) | Until 30 days after the last dose of the study drug
  Time to progression as assessed by the Investigator at local site per RECIST 1.1, or death due to any cause
Maximum plasma concentration (Cmax) | From pre-dose to 30 days after the last dose of the study drug
  Pharmacokinetic profile of NWY001
Time to Cmax (Tmax) | From pre-dose to 30 days after the last dose of the study drug
  Pharmacokinetic profile of NWY001
Area under the plasma concentration-time curve from 0 to infinity (AUC 0-inf) | From pre-dose to 30 days after the last dose of the study drug
  Pharmacokinetic profile of NWY001
Tumor necrosis factor-α (TNF-α) | From pre-dose to 30 days after the last dose of the study drug
  Pharmacodynamic profile of NWY001
Interleukin-6 (IL-6) | From pre-dose to 30 days after the last dose of the study drug
  Pharmacodynamic profile of NWY001
Incidence of anti-drug antibody (ADA) | From pre-dose to 30 days after the last dose of the study drug
  Immunogenicity of NWY001
Incidence of neutralizing antibody (NAb) | From pre-dose to 30 days after the last dose of the study drug
  Immunogenicity of NWY001

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, Ph.D., Principal Investigator — Sun Yat-sen University Cancer Cancer
Locations (1):
- Sun Yat-sen University Cancer Cancer, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No